CLINICAL TRIAL: NCT06751576
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Comparative Accuracy Of Readers Assisted By an AI/ML Technology-Based End-To-End CADe/CADx SaMD Versus Alone in the Detection, Localization and Characterization of Pulmonary Nodules in Populations With High Risk of Lung Cancer (RELIVE)
Brief Title: Retrospective Clinical Trial Comparing Radiologists' Diagnosis Accuracy in Lung Cancer Screening Population With and Without the Help of an AI/ML Tech-based SaMD
Acronym: RELIVE
Status: Completed | Type: Observational
Sponsor: Median Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MT-LCS-004
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: High Risk Cancer; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control arm: low-dose CT scan image readings performed by radiologists without the assistance of Median LCS
- Test arm: low-dose CT scan image readings performed by radiologists with the assistance of Median LCS.
  Interventions: Device: Median LCS

INTERVENTIONS:
Device: Median LCS — End-to-end processing of chest LDCT DICOM images by an AI/ML tech-based SaMD to detect, localize, and characterize (assign a malignancy score) each detected pulmonary nodule. The output of the device is a DICOM File (Median LCS result report) summarizing results per patient.
  Other Names: eyonis LCS
  Groups: Test arm

SUMMARY:
This is a two arm, randomized, controlled, blinded, multi-case multi reader (MRMC), retrospective study for the evaluation of the efficacy and safety of an AI/ML technology-based CADe/x developed to detect, localize and characterize malignancy score of pulmonary nodules on LDCT chest scans taken as part of a lung cancer screening program.

LDCT DICOM images of patients who underwent routine lung cancer screening will be selected and enrolled into the study. Enrolled scans analyzed by radiologists with the assistance of the Median LCS (formerly iBiopsy) device are compared to the analysis by radiologists without the assistance of the Median LCS device.

Figures of merit for patient level and lesion level detection and diagnostic efficacy will be calculated and compared, sub-class analysis will be performed to ensure device generalizability.

ELIGIBILITY:
Inclusion Criteria:

* ≥50-80 Years of age;
* Current or ex-smoker (>=20 pack years);
* Patient screened and surveilled for lung cancer screening following lung cancer screening guidelines (equivalent to United States Preventive Services Task Force (USPSTF) 2021 Criteria);
* Received LDCT due to inclusion in high-risk category for lung cancer.

Exclusion Criteria:

* Prior lung resection;
* Pacemaker or other indwelling metallic medical devices in the thorax that interfere with CT acquisition;
* Patients/images used during AI model development;
* Patients with only hilar and/or mediastinal cancer(s);
* Patients with only ground glass cancer(s);
* Patients with nodules, solid or part-solid >30mm (masses);
* Patients that are not accompanied with the required clinical information;
* Patients with imaging with any of the following: missing slices, slice thickness >3mm;
* Partial cover of the lung.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk lung cancer population from Radiology or Pneumology hospital departments.
  Patients enrolled in this study were retrospectively collected from centers across the EU and USA where they were enlisted into lung cancer screening due to high risk of lung cancer according to established lung cancer screening guidelines.
  The cohort used for testing the efficacy and safety of the device will be an "enriched cohort" with a 1:2 distribution of cancer positive and benign patients
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
∆ AUC of ROCs > 0. Delta Area between the Response operating curve (AUROC) value with Median LCS and AUROC without Median LCS at patient level data is superior to 0. | 12 months
  Demonstrate that patient diagnosis with Median LCS is improved compared to without Median LCS.

SECONDARY OUTCOMES:
Sensitivity at max Youden | 12 months
  Demonstrate that Median LCS aided sensitivity is non inferior (H2) , superior (H8) to radiologist alone.
  (Sensitivity with Median LCS-Patient) non inferior using non-inferiority margin delta = 0.1 to (Sensitivity Control Arm-Patient).
  First, non-inferiority. If passed, superiority will be performed.
Specificity at max Youden | 12 months
  Demonstrate that Median LCS assisted specificity is not inferior (H3), superior (H9) to radiologist alone.
  (Sensitivity with Median LCS-Patient) non inferior using non-inferiority margin delta = 0.1 to (Sensitivity Control Arm-Patient).
  First, non-inferiority. If passed, superiority will be performed.
∆ AUC of LROC > 0 | 12 months
  Demonstrate that Median LCS improves clinician's performance in finding detection and diagnosis.
Recall rates for non-cancer patients (Specificity) | 12 months
  Demonstrate that Median LCS aids to rule out non-cancer patients compared to radiologist alone.
  "Non-Cancer-Recall-Rate will be calculated and compared between the two modalities using margin of 10%". First, non-inferiority. If passed, superiority will be performed.
Recall rates for cancer patients (Sensitivity) | 12 months
  Demonstrate that Median LCS aid to diagnose cancer patients compared to radiologist alone.
  "Cancer-Recall-Rate will be calculated and compared between the two modalities using margin of 10%". First, non-inferiority. If passed, superiority will be performed.
Time analysis | 12 months
  Demonstrate that Median LCS decreases the time of analysis per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Anil VACHANI, MD, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (3):
  - University of Pennsylvania - Penn Center for Innovation, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Fundacion instituto de investigacion sanitaria de la fundacion jimenez diaz (FJD), Madrid
  - Universidad de Navarra, Pamplona